CLINICAL TRIAL: NCT01735851
Title: Comparison of Bilateral Thoracic Paravertebral Block to Thoracic Epidural Analgesia for Post Operative Analgesia in Patients Undergoing Abdominal Surgery - A Randomized Open Label Study
Brief Title: Comparison of Bilateral Thoracic Paravertebral Block to Thoracic Epidural Analgesia for Post Operative Analgesia in Patients Undergoing Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Sugantha Ganapathy, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSREB UWO 103035
Record Dates: First submitted 2012-10-26; First posted 2012-11-28 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Pain
Keywords: Thoracic epidural analgesia; Paravertebral block; pain; postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic epidural analgesia (Active Comparator): Group 1 will receive a catheter congruent TEA. The epidural space will be identified using the loss of resistance technique. After a test dose to rule out intravascular and intrathecal placement of the catheterthe initial block will be made with 0.25% bupivacaine 5 mL followed by 3 mL aliquots administered every 5 minutes to establish a block between T8 and T12. An infusion will be started at 8 mL/hour with 0.1 % bupivacaine with 10microgram/mL of dilaudid and continued for 72 hours. Additional nurse administered boluses of 5-10mL of the standard solution will be allowed via the epidural catheter every 6hourly for poor pain control followed by an increase in the basal infusion rate up to a maximum of 14mL/hr. Patients will be allowed to self administer additional boluses of 3mL of the standard infusate every 20minutes (PCEA)
  Interventions: Drug: Thoracic epidural analgesia
- Bilateral Paravertebral block (Experimental): Group 2 will have bilateral PVB catheters inserted using the ultrasound with patients prone. A high-frequency linear probe will used to visualize the transverse process, pleura and the internal intercostal membrane. A 17 guage Tuohy needle will be inserted to puncture the internal intercostal membrane. Injection of local anesthetic will push the pleura away, which will be the end point of needle position. A curved pigtail catheter will be inserted and further 5mL of local anesthetic will be injected while observing further movement of pleura. A similar procedure will be done on the contralateral side at the same level. Infusion of 0.2% ropivacaine will be continued for the next 72 hours. They will also receive IVPCA and additional nurse administered boluses of 5-10mL of ropivacaine 0.2% in the PVB every 6 hourly to the side of maximal pain.
  Interventions: Procedure: Bilateral Paravertebral block

INTERVENTIONS:
Drug: Thoracic epidural analgesia
  Other Names: Thoracic Epidural Anesthesia
  Arms: Thoracic epidural analgesia
Procedure: Bilateral Paravertebral block
  Arms: Bilateral Paravertebral block

SUMMARY:
Pain following abdominal surgery is managed with the use of thoracic epidural analgesia (TEA) where the epidural is inserted in the spine at the level of scapula The risks due to TEA include difficulty with insertion, failure in up to 40% of patient in the perioperative period, fall in blood pressure and a rare devastating complication of paralysis either due to bleeding or infection. Injury to spinal cord is also a feared complication. Therefore alternative techniques need to be evaluated. Paravertebral block (PVB) has been documented to provide pain relief following abdominal surgery using an earlier technique which posed the risk of puncture of the covering to the lung (pleura) resulting in pneumothorax. The current technique involves the use of curled catheters inserted using ultrasonography to lie outside the pleura where the nerves travel thus reducing the chances of pneumothorax and catheter migration. Objective of the current study is to compare the efficacy and safety of bilateral PVB with TEA. Patients undergoing bowel surgery will be randomized to receive thoracic epidural analgesia or bilateral thoracic paravertebral blocks. Pain scores during rest and coughing, failure and complication rates will be compared between the two groups.

Objective:

The objective of the investigators is to determine whether ultrasound (US)-guided bilateral thoracic paravertebral blocks (PVB) using curled catheter provides effective post-operative analgesia as compared to thoracic epidural analgesia in patients undergoing open abdominal bowel surgeries.

The primary outcome of this study will be the pain scores over the first 24 hours following open bowel surgeries.

Secondary outcomes include

1. Analgesic consumption in the perioperative period,
2. Block related data (block performance time, success rate, extent of sensory block, complications)
3. Hemodynamic parameter every 6 hourly
4. Incidence of side effects like nausea and pruritus scores, time to return of bowel activity

Hypothesis

Null Hypothesis: Primary.

Paravertebral blocks provide equal analgesia in the early postoperative period (first 24 hours of surgery) as compared to thoracic epidural analgesia in patients undergoing bowel surgeries by laparotomy.

Secondary

1. The analgesic consumption between PVB and TEA is not different during the first 24 hours following surgery
2. The block performance time, success rate and extent of sensory block with PVB are not different from that of TEA.
3. Side effects and complications following bilateral PVB are not different from those occurring after TEA

DETAILED DESCRIPTION:
A total of 70 patients with ASA physical status 1 to 3, scheduled for elective bowel surgery by laparotomy and deemed suitable to receive either thoracic paravertebral or epidural analgesia will be included in the study. Recruitment will take place in the preoperative clinic. Written informed consent for the participation in the study will be obtained at the visit to the preadmission clinic or in the preparation area at least 2 hours prior to the surgery. They will be randomized to one of two groups prior to the block procedure using a closed envelope system. All patients will be educated regarding the VRS scores on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain ever experienced. All patients will receive perioperative multimodal analgesia using naproxen, gabapentin and acetaminophen.

All blocks will be performed in the block room using standard monitoring, sterile precautions and titrated intravenous sedation with fentanyl and midazolam. During block performance one anesthetist and one assistant will be present. Due to the necessity of handling the equipment these staff will not be blinded. All patients will receive supplemental oxygen.

Group 1: Group 1 will receive a catheter congruent TEA. The catheters will be inserted using ultrasound to assess level as well as the best space to insert the epidural catheter between T7 and T9. The epidural space will be identified using the loss of resistance technique. After a test dose to rule out intravascular and intrathecal placement of the catheter using 3mL of 2% lidocaine with 5mcg/mL of epinephrine, the initial block will be made with 0.25% bupivacaine 5 mL followed by 3 mL aliquots administered every 5 minutes to establish a block between T8 and T12. An infusion will be started at 8 mL/hour with 0.1 % bupivacaine with 10 microgram/mL of dilaudid and continued for 72 hours. Additional nurse administered boluses of 5-10mL of the standard solution will be allowed via the epidural catheter every 6hourly if needed for pain control followed by an increase in the basal infusion rate up to a maximum of 14mL/hr. Patients will be allowed to self-administer additional boluses of 3mL of the standard infusate every 20minutes (PCEA) as per the standard practice at this hospital. Time to initiate the block and the failures will be documented. If the block fails, patients will receive intravenous PCA with dilaudid and the patient will be dropped out of the study for efficacy data.

Group 2 will have bilateral PVB catheters inserted using the ultrasound. Patients will be in prone position and will receive intravenous sedation similar to Group 1. The T8 spine will be identified and marked counting from the lumbar area. A high-frequency linear ultrasound probe will be positioned in the T8/9 intercostal space with the transverse process and pleura in the field as well as the internal intercostal membrane. (about 2.5 cm lateral to the spinous process) Using ultrasound guidance and an in-plane approach, a 17 gauge Tuohy needle connected to 15 mL of 0.5% ropivacaine via an extension tubing will be inserted to puncture the internal intercostal membrane. Injection of local anesthetic will push the pleura away, which will be the end point of needle position (the current standard technique in the the investigators institution). A curved pigtail catheter will be inserted while observing its delivery extrapleurally and further 5mL of local anesthetic will be injected while observing further movement of pleura. A similar procedure will be done on the contralateral side at the same level. The catheter will be secured to the skin and covered with dermabond and tegaderm. Following this, 0.2% ropivacaine will be infused at a rate of 7 mlLhr via each catheter for the next 72 hours post-operatively. They will also receive intravenous patient controlled analgesia with dilaudid at a dose of 0.2mg with a lock out of 6 mins. Additional nurse administered boluses of 5-10mL of ropivacaine 0.2% via the paravetebral catheters will be permitted every 6 hourly to the side of maximal pain. The position of the catheter will be confirmed on the routine post-operative chest x ray following the injection of contrast (Isovue: 2 mL). The sensory block extent will be documented at 15 minutes after the initial injection and prior to moving the patient to the OR. Time to initiate the block and the failure rate will be documented.

US image of paravertebral space before and after LA injection (IIM: internal intercostal membrane; TP: transverse process; LA: local anesthetic)

As soon as the arterial line is inserted in the operating room for monitoring purposes, 10mL of blood will be collected for measuring plasma ropivacaine levels. This measurement will be repeated on arrival in the PACU along with routine postoperative arterial blood gas analysis. Plasma ropivacaine level will be measured on postoperative day 1 at 6AM with the blood drawn along with routine postoperative blood work (venous sample)

Cases with a failure to establish a block 30 minutes after local anesthetic injection will be considered as block failure and the patient will be excluded from the efficacy part of the study. These patients will receive intravenous patient controlled analgesia. Once the effectiveness and level of the block is confirmed the patient will be moved to the operating room for the surgery under standardized general anesthesia using fentanyl 2-3µg/Kg, propofol 2 mg/kg and rocuronium 0.8-1.0 mg/kg for intubation followed by maintenance with desflurane in air-oxygen mixture. Vasopressors (Ephedrine and phenylephrine) will be administered as needed to control hemodynamics and the total dose used will be recorded.

The patients will be assessed for pain during rest and coughing/activity immediately after the surgery, every 15 minutes for first 2 hrs and 6 hourly thereafter until 24 hours after the removal of epidural or block catheters. Patients whose VRS scores are higher than 5/10 in PACU, apart from getting a bolus in the epidural or PVB may also receive IV Hydromorphone 0.2 mg every 5 minutes till pain subsides to a score of 3/10. Nausea will be documented using a categorical scale (none, mild, moderate and severe), pruritus scores will be recorded every 12 hours (categorical scale, none, mild, moderate and severe). Time to onset of bowel sounds, time to first flatus and time to first bowel movement would also be recorded with time 0 being the arrival time in PACU. Post-operative hemodynamic changes, blood pressure and urine output will be documented every 6 hours. Duration of significant hypotension will be computed from the nursing chart, significant hypotension being systolic BP less than 90 mm Hg. Patient satisfaction will be documented on a visual analogue scale where 0 is totally dissatisfied and 100 is totally satisfied. Adverse events such as local anesthetic toxicity, wound infection, dehiscence, urinary retention, cognitive dysfunction and neurological deficits will be prospectively collected. The failure rate of both the techniques and the number of attempts will also be recorded.

This is an open label study to document the effectiveness of bilateral PVB in bowel surgeries. The investigators plan to do a double blind study following the present study if the results are encouraging. The second concern is that 2 different local anesthetics are used for the 2 limbs but at equianalgesic concentrations for the infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females of 18-85years of age, scheduled to undergo open abdominal surgeries.
2. ASA Class I, II, III -

Exclusion Criteria:

1. Patients with associated significant cardiac and respiratory disease
2. Patients with coexisting hematological disorder or with deranged coagulation parameters.
3. Patients with pre-existing major organ dysfunction such as hepatic and renal failure.
4. Patients with anatomical deformity of spine
5. Psychiatric illnesses
6. Emergency surgery
7. Lack of informed consent.
8. Allergy to any of the drugs used in the study
9. Contraindications to epidural analgesia -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores at rest and on coughing in the first 24 postoperative hours | From arrival in PACU until 24 hours of arrival in the PACU
  Pain scores at rest and coughing will be documented every 15 minutes for the first 2 hours in PACU and thereafter every 6 hourly until the first 24 hours. Patients may receive intravenous dilaudid boluses in the PACU if the pain scores are greater than 5. patients will be receiving IVPCA or PCEA depending on the group allocation in the PACU. The total dose of narcotic used will be documented.

SECONDARY OUTCOMES:
total pain scores till 72 hours postoperatively | from arrival in PACU to 3rd postoperative day (72 hours)
  Pain scores at rest and coughing will be documented every 15 minutes for the first 2 hours in PACU and thereafter every 6 hourly until the block catheters are removed at 72 hours. Patients may receive intravenous dilaudid boluses if the pain scores are greater than 5. The total dose of narcotic used will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Finucane BT, Ganapathy S, Carli F, Pridham JN, Ong BY, Shukla RC, Kristoffersson AH, Huizar KM, Nevin K, Ahlen KG; Canadian Ropivacaine Research Group. Prolonged epidural infusions of ropivacaine (2 mg/mL) after colonic surgery: the impact of adding fentanyl. Anesth Analg. 2001 May;92(5):1276-85. doi: 10.1097/00000539-200105000-00038. PMID 11323362
- [Background] Luyet C, Meyer C, Herrmann G, Hatch GM, Ross S, Eichenberger U. Placement of coiled catheters into the paravertebral space. Anaesthesia. 2012 Mar;67(3):250-5. doi: 10.1111/j.1365-2044.2011.06988.x. PMID 22321080
- [Derived] Sondekoppam RV, Uppal V, Brookes J, Ganapathy S. Bilateral Thoracic Paravertebral Blocks Compared to Thoracic Epidural Analgesia After Midline Laparotomy: A Pragmatic Noninferiority Clinical Trial. Anesth Analg. 2019 Sep;129(3):855-863. doi: 10.1213/ANE.0000000000004219. PMID 31425230